CLINICAL TRIAL: NCT01943032
Title: Discordant Hormonal Status Between Primary Tumor and Axillary Lymph Node in Breast Cancer Patients.
Brief Title: Discordant Hormonal Status of Breast Cancer.
Status: Completed | Type: Observational
Sponsor: National Cancer Institute, Thailand (Other Government)
Responsible Party: Principal Investigator, AKANIST PIYAPANT, MD.,FRCST., MD.,FRCST. Surgical Oncologist., National Cancer Institute, Thailand
Other Study IDs: EC 196/2010
Record Dates: First submitted 2013-09-10; First posted 2013-09-16 (Estimated); Last update posted 2013-09-20 (Estimated); Status verified 2013-09

CONDITIONS: Malignant Neoplasm of Breast.
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — Paraffin embedded tissue blocks of primary breast tumor and axillary lymph nodes.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Primary Breast Tumor: Immunohistochemical staining of paraffin embedded tissue blocks of primary breast tumor for estrogen and progesterone receptors was performed.
- Axillary Lymph Nodes.: Immunohistochemical staining of paraffin embedded tissue blocks of axillary lymph nodes for estrogen and progesterone receptors was performed.

SUMMARY:
The purpose of this study is to determine discordant hormonal status of primary breast tumor and metastatic breast cancer cells at regional lymph nodes in node positive breast cancer patients.

DETAILED DESCRIPTION:
Hormonal status between primary breast tumor and axillary lymph node were analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer patients stage I,II and III with axillary lymph nodes metastasis.

Exclusion Criteria:

* Breast cancer patients stage I,II and III without axillary lymph nodes metastasis.

Ages: 25 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Breast Cancer Patients Stage I,II and III.
Sampling Method: Non-Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2011-04; Primary Completion 2011-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Association of hormonal status between primary breast tumor and axillary lymph nodes | Up to 1 year
  Association of estrogen and progesterone status between primary breast tumor and axillary lymph nodes was analyzed by using the χ2 test

CONTACTS AND LOCATIONS:
Overall Officials: AKANIST PIYAPANT, MD.,FRCST., Principal Investigator — National Cancer Institute, Thailand
Locations (1):
- National Cancer Institute, Thailand., Ratchathewi, Bangkok, Thailand

REFERENCES:
- [Background] Cristofanilli M, Budd GT, Ellis MJ, Stopeck A, Matera J, Miller MC, Reuben JM, Doyle GV, Allard WJ, Terstappen LW, Hayes DF. Circulating tumor cells, disease progression, and survival in metastatic breast cancer. N Engl J Med. 2004 Aug 19;351(8):781-91. doi: 10.1056/NEJMoa040766. PMID 15317891
- [Background] Cristofanilli M. The biological information obtainable from circulating tumor cells. Breast. 2009 Oct;18 Suppl 3:S38-40. doi: 10.1016/S0960-9776(09)70270-X. PMID 19914540